CLINICAL TRIAL: NCT00386386
Title: Enzymatically Augmented Subcutaneous Infusion (EASI) In Out-Of-Hospital Care
Brief Title: Recombinant Hyaluronidase in Out-of-Hospital Setting: The EASI Access Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Stephen THomas, MGH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hylenex1
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Mass Casualty Incident; Dehydration
Keywords: hydration; prehospital; mass casualty incident
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Subject receives two infusions: One by EASI Access and one by IV access, at different sites
  Interventions: Other: hypodermoclysis via recombinant hyaluronidase-facilitated subcutaneous infusion

INTERVENTIONS:
Other: hypodermoclysis via recombinant hyaluronidase-facilitated subcutaneous infusion — Above

SUMMARY:
The study's overarching aim is to determine whether Enzymatically Augmented Subcutaneous Infusion (EASI) can assist in out-of-hospital situations characterized by mismatch between need for, and ability to achieve, access to the vascular compartment. One mechanism for providing access to the vascular compartment, subcutaneous infusion, is facilitated by administration of hyaluronidase; the hyaluronidase hydrolyzes hyaluronan the major subcutaneous diffusion barrier. Hyaluronidase thus increases local dispersion and absorption of subcutaneously administered drugs and fluids.

The EASI Access study is intended to be the first out-of-hospital study assessing FDA-approved Chinese hamster ovary-derived recombinant hyaluronidase (the recombinant product is hereafter referred to by the shorter brand name, Hylenex). The EASI Access will test some fundamental principles and will facilitate design and implementation of follow-up investigations (e.g. extension of access to non-ALS providers). For example, we will attempt to show that EASI access is simple, effective, and has few or no downsides as compared to IV access.

DETAILED DESCRIPTION:
Background Challenges to IV access outside the hospital The out-of-hospital setting can pose myriad challenges to the provider attempting to gain access to the intravascular compartment. In an individual patient encounter, placement of an intravenous (IV) catheter may be hampered by anatomy (e.g. venous collapse in hypotension), positioning (e.g. entrapment), and environmental conditions such as lighting and vehicular motion. These problems may be compounded in situations where multiple patients simultaneously require expedited IV access. Therefore, both "host" (i.e. patient) and "environment" (i.e. physical setting) parameters can contribute to a mismatch between desire for, and ability to achieve, access to the intravascular compartment.

The aforementioned issues with IV line placement all make the assumption of presence of an operator with appropriate Advanced Life Support (ALS)-level training and credentials. Such may not be the case in a mass casualty incident (MCI) situation, or in a situation where initial responders are Basic Life Support (BLS) level. Thus, consideration of potential barriers to intravascular compartment access should include "personnel" as well as "host" and "environment" parameters.

Case for importance of access to intravascular compartment Is intravascular access really important? Assuming that an EMS system could fiat easy and widespread access to the intravascular compartment in an MCI or more routine ALS or BLS response, is there impact on outcome? Unfortunately, as is often the case with EMS interventions, there is little or no randomized controlled evidence addressing the issue - in fact, related literature on penetrating trauma suggests that prehospital fluid resuscitation may be deleterious. However, clinical practice as well as standard emergency medicine and trauma resuscitation teaching (such as the Advanced Cardiac Life Support course and the Advanced Trauma Life Support text) do emphasize importance of early fluid resuscitation for a variety of injuries and illnesses.1 In addition, literature addressing MCI situations (e.g. crush injuries) makes a strong case for the importance of fluid replacement.2 Besides opening an avenue for fluid replacement, catheter-based access to the intravascular compartment allows for reliable delivery of medications. For patients who are not tolerating po intake, or for those who otherwise stand to benefit from parenteral drug delivery, catheter-based access to the intravascular compartment allows for administration of repeated doses of a variety of drugs while avoiding multiple (often painful) injections. Once the catheter is placed (currently, in a vein), the access line is available to both initial and subsequent caregivers.

It is obvious that out-of-hospital caregivers may use the access line for administration of drugs in the (limited) prehospital pharmacopoeia, but it is equally true that pre-establishment of intravascular access saves a step on arrival to the next level of care. Practitioners in today's EDs currently benefit, in savings of nursing time, from not having to take time to establish IV access in patients transported to the hospital by ALS units. This helps both the individual patient with pre-established IV access, since ED staff can immediately administer time-critical drugs - including those not in the ALS armamentarium - and also aids the resource-taxed ED whose staff can execute duties other than starting IV lines. Furthermore, though there is no concrete supporting evidence, common wisdom holds that placement of a (smaller) IV line and fluid administration through that line, may facilitate subsequent placement of a larger IV line due to more fluid in the vascular compartment.

Thus, the balance of evidence from a variety of standpoints (outcomes research, accepted practice and teaching, logistics) supports an argument that ability to gain access to the intravascular compartment is an important priority for out-of-hospital care. Importantly, it should be noted that for "ED" one could substitute "triage tent" or other MCI-related care site since intravascular compartment access is of obvious import in MCI/disaster-type situations.

Potential role for EASI Mechanism of subcutaneous infusion Subcutaneously administered drugs and infusates must traverse an interstitial matrix to enter the vascular or lymphatic system. The interstitium's resistance to drug permeation can be envisioned as functioning like a three-dimensional filter through which drugs/infusates must pass. There are large molecules such as elastin and collagen inhabiting a matrix of hydrated gel-like glycosaminoglycans and proteoglycans. Among the glycosaminoglycans is hyaluronan, which contributes to the resistance of fluid flow through the interstitium. Though hyaluronan is found in lower concentration than collagen in the skin, it plays a disproportionately large role in resisting fluid movement.3 Hyaluronidase modifies connective tissue permeability via hydrolyzing hyaluronic acid, effecting a cleavage of the glucosaminidic bond between N-acetylglucosamine and glucuronic acid moieties. The cleavage results in a decrease in viscosity of the cellular cement and promotes diffusion of injected fluids, facilitating their absorption. The decrease in viscosity is reversed within 24 hours, due to the rapid inactivation of the hyaluronidase enzyme and also due to the rapid turnover rate of skin hyaluronan.4, 5 So-called "spreading agents," historically derived from animal extracts, have been used clinically to facilitate dispersion and absorption of other drugs for over 50 years.4 The extensive history of spreading agent use was relevant to the FDA review of the new recombinant enzyme. Based in part upon the longtime uses of (nonrecombinant) hyaluronidase, the FDA approval for Hylenex states the drug is: "Indicated as an adjuvant to increase the absorption and dispersion of other injected drugs, for hypodermoclysis, and as an adjunct in subcutaneous urography for improving resorption of radiopaque agents." Subcutaneous infusion instead of, or prior to, IV infusion

Out-of-hospital clinical scenarios vary widely. It is certainly true that not all EMS patients, or MCI patients, need an IV line. However, it is easy to think of out-of-hospital situations in which rapidly and easily placed intravascular access could be very helpful, and in which standard IV catheters may not be the (sole) solution. To name but a few examples, there could be a:

* Single-patient encounter where the IV line is difficult to place
* Multi-car motor vehicle crash (MVC) site attended by many BLS, but few ALS, providers
* Marathon medical support tent confronted with scores of volume-depleted individuals
* Building collapse (e.g. in an earthquake) with numerous victims in whom simultaneous and timely fluid replacement can stave off crush-mediated renal failure Standard texts such as the American College of Surgeons' Advanced Trauma Life Support note that the need for IV access is often present in cases where there is no ability to place an indwelling vascular catheter. The ATLS text points out that fluid resuscitation in clinically challenging environments (e.g. austere conditions, MCI situations) is often of sufficient criticality that, in the absence of IV access, hydration should be attempted through oral or rectal routes. As the ACS Committee on Trauma writes, oral hydration has obvious aspiration and absorption risks, and rectal clysis (as it is denoted in the ATLS text) presents obvious logistic and patient comfort issues in the field.1 It is thus clear that there is a potential role for EASI access if such access extends the ability to usefully reach the intravascular compartment. In terms of its potential as a mechanism for out-of-hospital fluid replacement and as a route for drug administration, EASI warrants attention in the form of a trial.

Compared to the current standard of IV (and perhaps intraosseous) line placement by ALS-level providers, EASI access could enable out-of-hospital responders (ALS as well as lower echelon providers) to achieve intravascular access in more patients, more quickly, more reliably, and with less pain. We thus plan to conduct the EASI Access study for out-of-hospital providers, as a mechanism to investigate whether EASI access can accrue the hypothesized advantages. The study will begin with ALS-level providers. The ultimate plan, should ALS provider EASI prove efficient, will be to assess whether simple placement of EASI access by non-ALS providers can extend the reach of advanced care providers in situations where need for IV access outstrips available resources.

Not specifically the goal of the EASI Access trial, but potentially relevant for any future use of Hylenex, is that the ability to avoid IV access may be occasionally useful in the acute care setting. In patients who are very young, or cachectic, or simply need IV access for fluid replacement, EASI may be able to obviate the need for (possibly numerous) IV "sticks" and their attendant discomfort. The low, but nonzero, rate of IV access complications (e.g. thrombosis, phlebitis) in general may also be avoided by use of EASI access. The EASI Access investigation very clearly does not offer these potential advantages to the current trial's study subjects, but the hypothetical advantages to avoiding IV placement do provide further possible relevance to any positive findings in the EASI Access study.

ELIGIBILITY:
Inclusion Criteria:

* Adults participating in disaster medicine drill

Exclusion Criteria:

* Diabetes
* Allergy to hyaluronidase or its components
* High doses of estrogens

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Ability to achieve hydration with subcutaneous infusion
Ability to get subcutaneously administered glucose into the vascular compartment
Safety of subcutaneous infusion
Rapidity of subcutaneous infusion as compared to standard IV infusion

SECONDARY OUTCOMES:
Pain associated with subcutaneous infusion vs. IV infusion

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Thomas, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Soremekun OA, Shear ML, Patel S, Kim GJ, Biddinger PD, Parry BA, Yialamas MA, Thomas SH. Rapid vascular glucose uptake via enzyme-assisted subcutaneous infusion: enzyme-assisted subcutaneous infusion access study. Am J Emerg Med. 2009 Nov;27(9):1072-80. doi: 10.1016/j.ajem.2008.08.028. PMID 19931753